CLINICAL TRIAL: NCT02840500
Title: Quality of Life Study in Patients With Cancer Breakthrough Pain Treated in Palliative Care Units
Acronym: CAVIDIOPAL
Status: Completed | Type: Observational
Sponsor: Angelini Farmacéutica (Industry)
Responsible Party: Sponsor
Other Study IDs: ANG-OPI-2016-01 (CAVIDIOPAL)
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Breakthrough Pain
Keywords: Breakthrough Cancer Pain; Quality of life; Palliative Care Units
MeSH Terms: conditions — Breakthrough Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breakthrough Cancer Pain: No intervention (Non-interventional study)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Patients treated in Palliative Care Units are potentially fragile patients, especially in our case, which are cancer patients. The management of these patients is usually done from experience, because these patients rarely meet criteria for clinical trials, as their inclusion could affect results obtained in the trial.

There is insufficient clinical information on the quality of life of cancer patients with breakthrough pain treated in palliative care units according to routine clinical practice. For this reason we consider it is appropriate to prospectively evaluate the quality of life of cancer patients with cancer breakthrough pain treated in palliative care units as well as the characteristics of these patients.

This post-authorization observational study will assess the quality of life of patients with breakthrough cancer pain treated in Palliative Care Units in Spanish hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* Patients with advanced cancer
* Patients attended in Palliative Care Units
* Life expectancy> 3 months
* Written informed consent
* Patients with baseline controlled cancer pain with opioids who are diagnosed of breakthrough cancer pain by Davies algorithm

Exclusion Criteria:

* Serious psychiatric disorder, cognitive impairment or any disease or condition that prevents the collection of data
* Patients with evidence of opioid addiction or history of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breakthrough cancer pain attended in Palliative Care Units will be included
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in quality of life according EORTC QLQ-C30 questionnaire | Baseline and 4 weeks
  Change in punctuation of the EORTC QLQ-C30 questionnaire between week 4 and baseline.

SECONDARY OUTCOMES:
Percentage of patients with neuropathic, visceral, somatic and mixed pain | Baseline (the day that patient sign the informed consent form)
  Percentage of patients with neuropathic, visceral, somatic and mixed pain
Comorbidities associated with patients | Baseline (the day that patient sign the informed consent form)
  Percentage of patients with each comorbidity
Change in mean Intensity of breakthrough cancer pain at each study visit | Up to 4 weeks, from date of inclusion until week 4
  Intensity of breakthrough cancer pain assessed with a Visual Analog Scale (VAS). VAS will be compared at each study visit.
Mean time to relief of breakthrough pain | Up to 4 weeks, from date of inclusion until week 4
  Time from the start of the episode until the relief of breakthrough pain
Mean duration of the episodes of breakthrough pain | Up to 4 weeks, from date of inclusion until week 4
  Time from the start of the episode until the pain ends
Patient Global improvement | Week 4
  Number of patients indicating each of the possible answers of the Patient Global Impression of improvement scale (7-points Likert scale)
Percentage of fragile patients at study entry | Baseline
  Frailty of patients will be assessed by Edmonton Symptom Assessment System (ESAS). It is considered that a patient is fragile when the symptom score is greater than 4 (moderate intensity) in five or more symptoms.
Cognitive impairment | Baseline
  Cognitive impairment (Pfeiffer test): 0-2 errors: intact cognition; 3-4 errors: mild impairment; 5-7 errors: moderate impairment; 8-10 errors: severe impairment. Percentage of patients in each category

CONTACTS AND LOCATIONS:
Overall Officials: Albert Tuca, MD, Study Director — Hospital Clinic de Barcelona, Palliative Care Unit
Locations (10):
- Spain (10):
  - Hospital de Mollet, Mollet del Vallès, Barcelona
  - Hospital Sant Joan de Deu, Palma, Illes Baleares
  - Hospital Clínic, Barcelona
  - Hospital Virgen de las Nieves, Granada
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Gregorio Marañón, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Complejo Hospitalario de Ourense, Ourense
  - Hospital Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez AT, Viejo MN, Maradey P, Canal-Sotelo J, Mancilla PG, Rivero SG, Casillas IR, Abian MH, Bermudo CL. Low-dose sublingual fentanyl improves quality of life in patients with breakthrough cancer pain in palliative care. Future Oncol. 2022 May;18(14):1717-1731. doi: 10.2217/fon-2021-1639. Epub 2022 Feb 9. PMID 35137627
- [Derived] Tuca Rodriguez A, Nunez Viejo M, Maradey P, Canal-Sotelo J, Guardia Mancilla P, Gutierrez Rivero S, Raja Casillas I, Herrera Abian M, Lopez Bermudo C. Impact of individualized management of breakthrough cancer pain on quality of life in advanced cancer patients: CAVIDIOPAL study. Support Care Cancer. 2021 Aug;29(8):4799-4807. doi: 10.1007/s00520-021-06006-1. Epub 2021 Feb 3. PMID 33533986